CLINICAL TRIAL: NCT02276976
Title: MRI,Gene And Cognitive Performance Study of Patients With Cerebral White Matter Lesions
Brief Title: MRI,Gene And Cognitive Performance Study of Patients With Cerebral White Matter Lesions(WMLs)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wei Wang (Other)
Responsible Party: Sponsor-Investigator, Wei Wang, professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: 2013BCB022
Record Dates: First submitted 2014-10-25; First posted 2014-10-28 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Cerebral White Matter Lesions
Keywords: crebral white matter lesions; brain networks; MRI; DTI; fMRI; cognitive impairment; gene
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- cerebral white matter lesions: patients with MRI confirmed cerebral white matter lesions
- healthy volunteers: healthy volunteers 1:1 matched by age,sex and education years

SUMMARY:
The purpose of this study is:1)to observe topological organization in brain structural and functional networks in cerebral white matter lesion patients and to evaluate the association between impairment of cognitive function and cerebral structural and functional networks in those patients;2)to indicate the role of genetic factors in the occurrence and prognosis of cerebral white matter lesions

DETAILED DESCRIPTION:
100 patients with cerebral white matter lesions and 100 normal controls will be observed. All of them will receive MRI scan(T1WI,T2WI,T2flair,MRA,SWI,ASL,DTI and fMRI) and the assessment of the neuropsychological function (MMSE,Auditory verbal memory test,Trail-making test-A and -B,Symbol digit modalities test,Digit span test,Clock drawing test,HAMD) intending to analyse topological organization in brain structural and functional networks in cerebral white matter lesion patients and to evaluate the association between impairment of cognitive function and cerebral structural and functional networks in those patients.Furthermore,DNA will be extracted from the blood sample of all participates to perform High-throughput sequencing. MRI scan and neuropsychological function assessment will be performed repeatedly after 1,3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* MRI diagnosis of cerebral white matter lesions Must be able to measure his(her) neuropsychologic function No severe stroke history and no physical disability Patients aged 40 to 85 Based on China's relevant laws, the patient himself agreed to participate in this study, a good compliance.Patients himself/herself must sign informed consent moreover

Exclusion Criteria:

* Unable to undergo examinations due to disturbances of consciousness or medical conditions Serious complications including severe heart failure, hepatic dysfunction, renal insufficiency,or shock AD,Parkinson's disease, malignant tumor, MS and other autoimmune diseases toxic and metabolic encephalopathy cerebral white matter lesions caused by CADASIL and other confirmed monogenic disease

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with cerebral white matter lesions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
MRI and cognitive function scale | up to 5 years after first assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Neurology of Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China